CLINICAL TRIAL: NCT02226757
Title: Paclitaxel-trastuzumab in EGFR-mutated NSCLC Patients After Progression on TKI-treatment; a Pilot-study
Brief Title: Paclitaxel-trastuzumab in EGFR-mutated NSCLC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof. dr. E.F. Smit, MD PhD, Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HER2-targeting in EGFR-mutated
Record Dates: First submitted 2014-06-02; First posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: NSCLC; HER2-expression; EGFR-mutation
Keywords: NSCLC; HER2-expression; EGFR-mutation; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel-trastuzumab (Experimental): Paclitaxel-trastuzumab weekly
  Interventions: Drug: Paclitaxel-trastzumab

INTERVENTIONS:
Drug: Paclitaxel-trastzumab — Trastuzumab
  * Dose:
    * First dose: 4 mg/kg IV
    * Subsequent doses: 2 mg/kg every week IV.
  * The patient must be monitored for at least 6 hours after the start of the first infusion and for at least 2 hours after the start of subsequent infusions.
  Paclitaxel
  - Dose: 60 mg/m2 IV in 30 minutes, every week, after trastuzumab

SUMMARY:
This study is a pilot study in EGFR-mutated NSCLC patients who have progressed on standard-dose TKIs. Tumor biopsies will be evaluated for HER2-expression. In case of HER2 expression, patients can participate in the trial after obtaining informed consent.

Patients will be treated with weekly paclitaxel-trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV non-squamous NSCLC patients.
* Patients must have been detected with an activating EGFR mutation at baseline and must have yet progressed on erlotinib, gefitinib or afatinib monotherapy in daily dose of 150 mg, 250 mg or 40 mg respectively. (Patients with unknown mutation status that have exhibited a response to these agents or stable disease for at least 6 months while on treatment with gefitinib or erlotinib are also eligible).
* Rebiopsy after having acquired resistance to TKI-treatment must have been performed and HER2-overexpression (positive immunohistochemistry staining) must have been detected.
* There must be at least one measurable disease site, according to RECIST 1.1 criteria.
* WHO performance status 0-2.
* Willing and able to comply with the study prescriptions.
* 18 years or older.
* Not pregnant or breast feeding and willing to take adequate contraceptive measures during the study.
* Ability to give written informed consent before patient registration.

Exclusion Criteria:

* No uncontrolled infectious disease.
* No other active malignancy.
* No major surgery (excluding diagnostic procedures like e.g. mediastinoscopy or VATS biopsy) in the previous 4 weeks.
* No treatment with investigational drugs.
* No known hypersensitivity to trastuzumab-paclitaxel
* No symptomatic brain metastases.
* History of coronary artery disease, NYHA class III or IV and Left Ventricular Ejection Fraction (LVEF) of <45%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 weeks

SECONDARY OUTCOMES:
Disease control rate | 6 weeks
progression-free survival | 2 years
Toxicity | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- VU University medical Center, Amsterdam, Netherlands